CLINICAL TRIAL: NCT03014765
Title: Endothelial Dysfunction, Indicator of Perioperative Complications and Its Changes in Perioperative Period
Brief Title: Endothelial Dysfunction in Perioperative Period
Acronym: EDOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Loyola University (Other)
Responsible Party: Principal Investigator, Peter Poredos, Head of Orthopaedic Anaesthesia, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MZ 0120-446/2015-2
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Endothelial Dysfunction; Postoperative Complications
Keywords: endothelial dysfunction; perioperative stress; cardiovascular complications; inflammatory markers
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: EDOP — no intervention

SUMMARY:
Study will enroll patients scheduled for hip arthroplasty. In each subject a flow-mediated dilatation capability (FMD) of the brachial artery will be measured prior to elective surgery, within 24 hours after surgery and 5-7 days after surgery. At each session the brachial artery diameter will be measured at rest, during cuff inflation and 50 seconds after cuff deflation. From above mentioned values the increase in the diameter of the artery during reactive hyperemia will be calculated.

Simultaneously with the ultrasound investigations, the blood for determination of the endothelial dysfunction markers will be collected.

The participants will be contacted again 3 months after the surgery and asked about the complications which may be associated with the surgery.

DETAILED DESCRIPTION:
Cardiovascular complications, especially coronary heart disease, are one of the main causes of perioperative complications. Indicators of pre-clinical atherosclerosis, such as: endothelial dysfunction, increased arterial intima/media thickness (especially in the carotid arteries), carotid calcification and coronary calcification, suggest the presence of atherosclerotic process without the symptomatic presentation. Endothelial dysfunction is one of the earliest measurable changes that predict the development of atherosclerotic disease.

Surgery is a significant stress for the organism: it increases the release of free oxygen radicals and through oxidative stress it increases systemic inflammatory response and causes thromboembolic complications.

In the study 50 patients of both sexes 40-80 years of age scheduled for hip arthroplasty will be included. In each subject a flow-mediated dilatation capability (FMD) of the brachial artery will be measured prior to elective surgery, within 24 hours after surgery and 5-7 days after surgery. Measurement of the brachial artery flow-mediated dilatation capability (FMD): the brachial artery diameter will be measured 5 cm proximal to the antecubital fossa at rest, during cuff inflation and 50 seconds after cuff deflation. The cuff will be inflated for 4 min. From above mentioned values the increase in the diameter of the artery during reactive hyperemia will be calculated.

Simultaneously with the ultrasound investigations, the blood for determination of the inflammatory and endothelial dysfunction markers (CRP, IL-6, IL-8, IL-10, IL-18, TNFa, VW Factor, Selectin P, selectin E) will be collected.

The participants will be contacted again 3 months after the surgery and asked about the complications which may be associated with the surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled hip arthroplasty under spinal anesthesia

Exclusion Criteria:

* Acute coronary syndrome or cerebrovascular syndrome in the last 6 months
* Acute venous thrombosis in the last 6 months
* Episode of rheumatoid arthritis in the last 3 months or permanent therapy with prednisolone >4mg/day
* Acute illness or hospitalization in the last month
* Chronic kidney failure on dialysis
* Hepatic failure
* Active malignant disease
* Immunosuppression after organ transplantation
* Pregnancy
* No informed consent after oral and written information

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
rate of perioperative cardiovascular complications in patients scheduled for hip arthroplasty under spinal anesthesia related to endothelial dysfunction | 12 months

SECONDARY OUTCOMES:
levels of blood circulating markers of increased perioperative stress and systemic inflammatory response | 12 months
  levels of vWF, selectin P, selectin E, IL-6, IL-8, IL-10, IL-18, TNFa
decrease in endothelial function | 12 months
  reduction in dilatation capability of brachial artery in the perioperative period - the difference between preoperative and postoperative values

IPD SHARING:
Plan to Share IPD: No